CLINICAL TRIAL: NCT07065630
Title: A Phase II Study of Volrustomig, Paclitaxel, and Carboplatin Followed by Response-Adaptive Treatment in Untreated Locoregional HPV-Negative Head and Neck Cancer
Brief Title: Response-Adaptive Treatment in Untreated Locoregional HPV-Negative Head and Neck Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-0567
Record Dates: First submitted 2025-06-02; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; HPV
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Volrustomig (Experimental): Dose Level 0: 500 mg IV on day 1 of 21-day cycle Dose Level 1: 750 mg IV on day 1 of 21-day cycle
  After the completion of radiation, patients will be initiated on maintenance volrustomig. Volrustomig will be administered at 250mg on day 1 of a 21-day cycle for 12 cycles (36 weeks/9 months)
  Interventions: Drug: Volrustomig
- Carboplatin (AUC) (Experimental): Dose Level 0: AUC 5 IV on day 1 of 21-day cycle Dose Level 1: AUC 5 IV on day 1 of 21-day cycle
  Interventions: Drug: Carboplatin
- Paclitaxel (mg/m2) (Experimental): Dose Level 0: 100 mg/m2 IV on Day 1 and Day 8 of 21-day cycle Dose Level 1: 100 mg/m2 IV on Day 1 and Day 8 of 21-day cycle
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Volrustomig — 500mg or 750mg (cycles 1-2) and 250mg thereafter IV day 1.
  Arms: Volrustomig
Drug: Carboplatin — 100mg/m2 IV day 1 and day 8.
  Arms: Carboplatin (AUC)
Drug: Paclitaxel — AUC 5 IV day 1
  Arms: Paclitaxel (mg/m2)

SUMMARY:
The purpose of this study is to assess the objective response rate following neoadjuvant therapy with volrustomig, paclitaxel, and carboplatin in previously untreated human papillomavirus (HPV)-negative locally advanced head and neck squamous cell carcinoma

.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed locally advanced, non-metastatic, head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, nasopharynx, larynx, or sinuses.

  * If a primary oropharyngeal squamous cell carcinoma is diagnosed, HPV must be ruled out by immunohistochemistry (defined as negative immunohistochemical staining of p16)
  * Non-oropharyngeal primary sites do not require immunohistochemical or other means of testing for HPV status, however if they are performed, must be negative for HPV.
  * Nasopharyngeal primary must have both EBV and HPV ruled out by immunohistochemistry to be eligible.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Stage IV disease with the exception of nasopharyngeal primary T3N2 (stage III) based of AJCC staging 8th edition.
* Patients must have measurable disease per RECIST 1.1 criteria, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* No previous radiation, chemotherapy, or immunotherapy for a head and neck cancer.
* Age ≥18 years.
* ECOG performance status of 0 or 1.
* Patients must have adequate organ and marrow function as defined below

  * Leukocytes ≥3,000/mcL
  * Absolute neutrophil count ≥ 1.5 × 109/L (1,500 per mm3)
  * Platelet count ≥ 100 × 109/L (100,000 per mm3)
  * Hemoglobin ≥ 9.0 g/dL (5.59 mmol/L)
  * Total bilirubin ≤ 1.5 × ULN in the absence Gilbert's syndrome ≤ 3×ULN if the subject has Gilbert's syndrome
  * Alanine transaminase and aspartate transaminase ≤ 3 × ULN
  * LVEF as assessed by echocardiography or multiple-gated acquisition scan ≥ 50%
  * Troponin I or T≤ ULN (institutional guidelines and/or not clinically significant per investigator judgement)
  * QTcF ≤ 480 msec
  * Creatinine within normal institutional limits OR eGFR (using CKD-EPI equation)≥45 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* No complete surgical resection for a head and neck cancer within 8 weeks of enrollment (although lymph node biopsy including excision of an individual node with presence of residual nodal disease, or surgical biopsy/excision of the tumor with residual measurable disease is acceptable.) No surgical procedures will occur after baseline scans are performed and measurable lesions are identified, although fine needle aspiration or core needle biopsies can be performed without need to repeat baseline scans before starting treatment if otherwise within screening window.
* The effects of volrustomig on the developing human fetus are unknown. For this reason and because anti-PD1/anti-CTLA4 agents as well as other therapeutic agents used in this study are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of volrustomig administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Unequivocal demonstration of distant metastatic disease (M1 disease).
* Unidentifiable primary site.
* Prior surgical therapy other than incisional/excisional biopsy or organ-sparing procedures such as debulking of airway-compromising tumors. Residual measurable tumor is required for enrollment as discussed above.
* Patients who are receiving any other investigational agents.
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are free of disease for ≥ 3 years. Exceptions include other cancers that have undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence life expectancy in the subsequent 3 years without active treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to volrustomig or other agents used in study.
* Patients with uncontrolled intercurrent illness.
* Negative pregnancy test (urine or serum) for female subjects of childbearing potential. Female subjects must be 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception (an acceptable method of contraception is defined as a barrier method in conjunction with a spermicide) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of volrustomig to prevent pregnancy. In addition, oral contraceptives, approved contraceptive implant, long-term injectable contraception, intrauterine device, or tubal ligation are allowed. Oral contraception alone is not acceptable; additional barrier methods in conjunction with spermicide must be used. Pregnant women are excluded from this study because volrustomig is an anti-PD1/anti-CTLA4 agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with volrustomig, breastfeeding should be discontinued if the mother is treated with volrustomig. These potential risks may also apply to other agents used in this study.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of Volrustomig monotherapy.
* Male subjects must be surgically sterile or using an acceptable method of contraception (defined as barrier methods in conjunction with spermicides) for the duration of the study (from the time they sign consent) and for 3 months after the last dose of Volrustomig to prevent pregnancy in a partner.
* Intercurrent medical illnesses which would impair patient tolerance to therapy or limit survival. This includes but is not limited to ongoing or active infection, immunodeficiency, specified cardiac conditions (below), pulmonary dysfunction, cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance. Patients with clinically stable and/or chronically managed medical illnesses that are not symptomatic and/or are not expected to impact treatment on protocol are still eligible.
* Any of the following cardiac conditions:

  * Cardiomyopathy of any etiology or history of myocarditis
  * Heart failure (as defined by New York Heart Association class III-IV)
  * Uncontrolled hypertension
  * Unstable angina pectoris
  * Clinically significant coronary, carotid, or peripheral artery stenosis
  * Acute coronary syndrome/acute myocardial infarction and/or coronary intervention with PCI/CABG within 12 months prior to randomization
  * Prior arterial or peripheral vascular intervention within 12 months prior to randomization
  * Ventricular arrhythmias requiring treatment, high degree AV block (II-III), or sinus node dysfunction with significant sinus pause, untreated with pacemaker. Note: Patients with atrial fibrillation or flutter who are clinically stable and have an optimally controlled ventricular rate (eg, mean of < 100 bpm on resting ECG or 24-h Holter-ECG) may be eligible if all other cardiac eligibility criteria are met, and a cardiology assessment confirms suitability for study treatment.
  * History of QT prolongation associated with other medications that required discontinuation of that medication.
  * Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives.
  * Planned or scheduled cardiac surgery or percutaneous coronary intervention procedure.
  * Planned revascularization procedure within 6 months of randomization.
* Evidence of the following infections:

  * Active infection including tuberculosis (TB) (clinical evaluation that includes clinical history, physical examination, and radiographic findings and TB testing in line with local practice).
  * Uncontrolled human immunodeficiency virus (HIV) infection; the following criteria are required to define well-controlled HIV infection:
  * undetectable viral RNA load for 6 months, CD4+ count of >500 cells/μL, stable for at least 6 months on the same anti-HIV medications, and no history of AIDS (defined by either CD+T cell count <200 cells/μL and/or AIDS-defining opportunistic infection)
  * Active or uncontrolled hepatitis B (HBV) or hepatitis C (HCV); Participants are eligible if they:
  * Have controlled hepatitis C viral load defined as undetectable hepatitis C RNA by PCR either spontaneously or in response to a successful prior course of anti-hepatitis C therapy
  * Have received HBV vaccination with only anti-HBs positivity and no clinical signs of hepatitis
  * Are HBsAg negative and anti-HBc+ (ie, those who have cleared HBV after infection) and meet conditions i-iii below:
  * Are HBsAg positive with chronic HBV infection (lasting 6 months or longer) and meet conditions i-iii below:
  * HBV DNA viral load <100 IU/mL
  * Have normal transaminase values Start or maintain antiviral treatment if clinically indicated as per the investigator. These patients will receive repeat testing at least every 6 months to assess for reactivation.
  * Active hepatitis A
* Diagnosis of immunodeficiency or is receiving systemic steroid therapy in excess of physiologic dose or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment.

The following are exceptions to this criterion:

* Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
* Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
* Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

  -Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years may be included but only after consultation with the study physician
* Patients with celiac disease controlled by diet alone.

  * History of allogenic organ transplantation.
  * Has known history of, or any evidence of active, non-infectious pneumonitis.
  * Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 90 days after the last dose of IP.
  * Subjects who are blood donors should not donate blood during the study and for 3 months following their last dose of volrustomig.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-17 (Estimated); Primary Completion 2029-08-13 (Estimated); Study Completion 2029-08-13 (Estimated)

PRIMARY OUTCOMES:
Response rate | 24 months
  Assess the objective response rate following neoadjuvant therapy with volrustomig, paclitaxel, and carboplatin in previously untreated human papillomavirus (HPV)-negative locally advanced head and neck squamous cell carcinoma (LA-HNSCC).
  The proportion of patients who achieve an objective response (30% or greater tumor shrinkage per RECIST v1.1 criteria) after chemoimmunotherapy.

SECONDARY OUTCOMES:
Survival outcomes | 24 months
  Assess in patients receiving neoadjuvant therapy with volrustomig, paclitaxel, and carboplatin followed by response-adaptive treatment in previously untreated HPV(-) LA-HNSCC.
  * Progression-free survival at 24 months.
  * Overall survival at 24 months.
Control of treatment failure | 24 months
  Assess disease control of treatment failure in patients receiving neoadjuvant volrustomig, paclitaxel, and carboplatin followed by response-adaptive treatment in previously untreated HPV(-) LA-HNSCC, and compare disease control and patterns of treatment failure between treatment arms.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 24 months
  Assess optimal dose and safety and tolerability of neoadjuvant volrustomig, paclitaxel, and carboplatin followed by response-adaptive treatment in previously untreated HPV(-) LA-HNSCC. Acute toxicity as assessed by CTCAE v5.0 measuring during treatment
Patterns of treatment failure | 24 months
  Assess disease patterns of treatment failure in patients receiving neoadjuvant volrustomig, paclitaxel, and carboplatin followed by response-adaptive treatment in previously untreated HPV(-) LA-HNSCC, and compare disease control and patterns of treatment failure between treatment arms.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States